CLINICAL TRIAL: NCT02528500
Title: Early Feasibility Assessment of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis in the Treatment of Type IV Thoracoabdominal Aortic Aneurysms Involving the Visceral Branch Vessels
Brief Title: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis in the Treatment of Type IV Thoracoabdominal Aortic Aneurysms
Acronym: TAMBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAA 13-02
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TAMBE Device (Experimental): Study designed to assess the feasibility of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device) in the treatment of patients with aortic aneurysms involving the visceral branch vessels. Patients with thoracoabdominal or pararenal abdominal aortic aneurysms are eligible for screening for participation in the study. The particular characteristics of the patient's aneurysm and anatomy will determine ultimate eligibility for enrollment. Only patients who meet all of the eligibility criteria will be enrolled.
  Interventions: Device: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis — Non-randomized, multicenter study designed to assess the initial feasibility of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device)
  Other Names: TAMBE Device

SUMMARY:
This study will assess the initial feasibility of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device) in the treatment of Aortic Aneurysms Involving the Visceral Branch Vessels.

DETAILED DESCRIPTION:
This is a prospective, non-randomized study designed to assess the feasibility of the TAMBE Device in the treatment of patients with aortic aneurysms involving the visceral branch vessels. A maximum of 10 Subjects will be treated under this Protocol. This clinical study will include up to six sites in the US. Each enrolled subject will undergo periodic follow-up evaluations involving physical exams, contrast-enhanced computed tomography (CT) of chest, abdomen and pelvis, creatinine measurement, abdominal ultrasound (optional) at specific, protocol-defined intervals for a period of five years following the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis implant.

ELIGIBILITY:
Inclusion Criteria:

1. Aortic aneurysm involving the visceral vessels requiring treatment
2. Adequate access for TAMBE Device components
3. Appropriate aortic anatomy to receive the TAMBE Device
4. Age ≥ 18 years at the time of informed consent signature
5. Male or infertile female
6. The patient is considered high risk for open repair as deemed by the treating physician
7. Capable of complying with protocol requirements, including follow-up
8. An Informed Consent Form signed by Subject or legal representative Note: Additional Inclusion Criteria may apply

Exclusion Criteria:

1. Prior aortic surgery
2. Ruptured or leaking aortic aneurysm
3. Aneurysmal dilatation due to chronic aortic dissection
4. Infected aorta
5. Mycotic aneurysm
6. Life expectancy <2 years
7. Myocardial infarction or stroke within 6 weeks of treatment
8. Systemic infection which may increase risk of endovascular graft infection
9. Degenerative connective tissue disease, e.g. Marfan's or Ehler-Danlos Syndrome
10. Participation in another drug or medical device study within 1 year of study enrollment
11. History of drug abuse, e.g. cocaine or amphetamine or alcohol, within 1 year of treatment
12. Tortuous or stenotic iliac and / or femoral arteries and the inability to use a conduit for vascular access
13. Known sensitivities or allergies to the device materials
14. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin
15. Patient has body habitus or other medical condition which prevents adequate fluoroscopic and CT visualization of the aorta
16. Renal Insufficiency Note: Additional Exclusion Criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2023-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Makaroun, M.D., Principal Investigator — University of Pittsburgh
Locations (6):
- United States (6):
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Mount Sinai Medical Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - UPMC, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Oderich GS, Farber MA, Silveira PG, Tadros R, Marin M, Fillinger M, Makaroun M, Hemmer J, Madden M. Technical aspects and 30-day outcomes of the prospective early feasibility study of the GORE EXCLUDER Thoracoabdominal Branched Endoprosthesis (TAMBE) to treat pararenal and extent IV thoracoabdominal aortic aneurysms. J Vasc Surg. 2019 Aug;70(2):358-368.e6. doi: 10.1016/j.jvs.2018.10.103. Epub 2019 Jan 3. PMID 30612825

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAMBE Device
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TAMBE Device
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 174.1 (9.72)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 86.4 (20.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (5.07)

OUTCOME MEASURES:

1. Primary Outcome: Absence of the Following Procedural Safety Events: Death, Stroke, Myocardial Infarction, Bowel Ischemia, Paraplegia, Respiratory Failure, Renal Failure, Procedural Blood Loss ≥1000 mL
Description: Absence of the following procedural safety events through 30 days post-procedure: Death, Stroke, Myocardial Infarction, Bowel Ischemia, Paraplegia, Respiratory Failure, Renal Failure, Procedural Blood Loss ≥1000 mL
Time Frame: Absence of procedural safety events through 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TAMBE Device
Number analyzed (Participants) | 10
Participants | 9

2. Secondary Outcome: Technical Success, Including Individual Components of Technical Success
Description: Components of Technical Success: Successful access to the necessary arterial sites, successful deployment of all required TAMBE Device components, Patency of all required TAMBE Device components and any required accessory components on completion angiography, absence of surgical conversion within 24 hours of initial of procedure
Time Frame: 12-month
Measure: Count of Participants; unit: Participants
Arm/Group | TAMBE Device
Number analyzed (Participants) | 10
Participants
  Technical Success | 9
  Successful Access | 10
  Successful Deployment | 10
  Patency of all required TAMBE Device components | 9
  Absence of Surgical Conversion | 10

3. Secondary Outcome: Device Integrity, Including Individual Components of Device Integrity
Description: Components of Device Integrity: Loss of functional patency in any treated branch component due to thrombus or mechanical failure of branch component, loss of functional patency in main body component(s) due to thrombus or mechanical failure of main body components(s) , separation of treated branch component from the main body component(s), separation of the main body component(s) from the accessory components
Time Frame: 12-month
Measure: Count of Participants; unit: Participants
Arm/Group | TAMBE Device
Number analyzed (Participants) | 10
Participants
  Loss of Functional Patency (Through 12M) | 2
  Separation of Components (Through 12M) | 0

4. Secondary Outcome: Patency (Primary, Assisted Primary, and Secondary)
Description: Primary Patency - Blood flow without occlusion maintained through the device without an intervention. Assisted Primary Patency: Blood flow maintained through the device after implant regardless of re-interventions performed. Secondary Patency - Blood flow through the device (following occlusion) regardless of re-interventions performed and freedom from surgical bypass.
Time Frame: 12-month
Measure: Count of Participants; unit: Participants
Arm/Group | TAMBE Device
Number analyzed (Participants) | 10
Participants
  Primary Patency (Through 12 Months) | 8
  Assisted Primary Patency (Through 12 Months) | 8
  Secondary Patency (Through 12 Months) | 9

5. Secondary Outcome: Absence of Type I and Type III Endoleaks at One Month Follow-up
Description: Absence of Type I and Type III endoleaks
Time Frame: One Month followup
Population: Includes only subjects with evaluable imaging within the one month window
Measure: Count of Participants; unit: Participants
Arm/Group | TAMBE Device
Number analyzed (Participants) | 8
Participants
  Absence of Type I Endoleak | 8
  Absence of Type III Endoleak | 8

ADVERSE EVENTS:
Time Frame: 5 Years
Arm/Group | TAMBE Device
All-Cause Mortality (participants affected / at risk) | 5/10
Serious Adverse Events (participants affected / at risk) | 10/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAMBE Device (N=10)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Illeus (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1)
Vascular stent stenosis (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1)
Cystilis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Squamos cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Spinal claudication (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Artery dissection (Vascular disorders) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAMBE Device (N=10)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ventricular dyssynchrony (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 2 (3)
Vascular stent occlusion (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal atrophy (Renal and urinary disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator agree not to submit any Publication until Study Completion and multi-center Publication has been published. If the multi-center Publication has not been submitted within 12 months of Study Completion, Institution and investigator may proceed with submission of the Publication; subject to the following: Investigator will provide all Publications to Sponsor for review that is more than 60 days but may extend an additional 120 days.

DOCUMENTS (2):
  • Study Protocol (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT02528500/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02528500/SAP_001.pdf